CLINICAL TRIAL: NCT03819842
Title: Evaluating the Need for Pseudophakic Intraoperative Abberrometry in Toric IOL Implantation
Brief Title: Evaluating the Need for the Pseudophakic Intraoperative Abberrometry in Toric IOL Implantation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alterman, Modi, & Wolter Ophthalmic Physicians & Surgeons (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: SSM--2017-12
Record Dates: First submitted 2019-01-22; First posted 2019-01-29 (Actual); Last update posted 2022-01-20 (Actual); Status verified 2022-01

CONDITIONS: Cataract; Nuclear Sclerosis; Cortical Cataract; Posterior Subcapsular Cataract; Astigmatism
Keywords: cataract surgery; cataract; toric IOL
MeSH Terms: conditions — Cataract; Astigmatism

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Aphakic Measure only (No Intervention): Eye measured in aphakic state only
- Pseudophakic measure (Active Comparator): Eye measured in aphakic state then again in pseudophakic state with toric IOL using the ORA System. Pseudophakic measurement obtained will provide data about placement of toric iol and the surgeon will use that data to rotate the iol if necessary.
  Interventions: Diagnostic Test: Pseudophakic Measurement

INTERVENTIONS:
Diagnostic Test: Pseudophakic Measurement — standard aphakic measurements will be taken and then pseudophakic measurements will be taken after toric iol implantation. The data produced will aid the surgeon in proper placement of toric iol orientation
  Arms: Pseudophakic measure

SUMMARY:
To determine clinically significant difference in results obtained from cataract surgery using IA. One eye will receive aphakic measurements only and the fellow eye will receive aphakic and then pseudophakic measurements when implanting a toric IOL.

DETAILED DESCRIPTION:
To determine if there is a clinically significant difference in the results obtained for the toric IOL implantation when using IA to measure the aphakic eye only and when using IA to measure the aphakic eye and then the pseudophakic eye, with toric IOL implantation.

ELIGIBILITY:
Inclusion Criteria:

* willing and able to understand and sign an informed consent
* willing and able to attend all study visits
* presenting for uncomplicated bilateral cataract surgery and have an interest in a toric iol
* have good ocular health, with no pathology that compromises visual acuity (outside of residual refractive error)
* have visually significant cataracts
* have regular corneal astigmatism of 1.0D to 5.0D in both eyes with a difference between eyes of 1.0D or less
* have potential post operative acuity of 20/25 or better

Exclusion Criteria:

* corneal pathology
* amblyopia
* prior corneal refractive surgery or other refractive surgery
* previous anterior or posterior chamber surgery that the investigator feels may compromise visual outcomes
* Diabetic retinopathy if the investigator feels this will compromise visual outcomes
* macular degeneration
* history of retinal detachment
* irregular astigmatism or keratoconus
* strabismus
* if in the surgeon's opinion the subject is not an appropriate candidate for iol implantation
* subjects who have an acute or chronic disease or illness that would confound the results of this investigation

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-03-19 (Actual); Primary Completion 2019-01-14 (Actual); Study Completion 2019-01-14 (Actual)

PRIMARY OUTCOMES:
Clinically significant difference in results obtained for tori iol implantation when using IA | 30 days
  Difference in magnitude of residual refractive astigmatism between groups Percentage of eyes with 0.50D or less of postoperative residual refractive astigmatism at 1 month post-op in each sub-group
  * Percentage of eyes within 0.50D of intended spherical equivalent
  * Sub-group analysis:
    * Vector analysis of the effects of any toric IOL realignment suggested by pseudophakic IA (i.e. was it likely to improve or worsen residual refractive astigmatism and/or UCVA)

CONTACTS AND LOCATIONS:
Locations (1):
- Alterman Modi and Wolter Ophthalmic Physicians and Surgeons, Poughkeepsie, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided
Results of the study may be shared at international meetings and submitted for peer review